CLINICAL TRIAL: NCT00572234
Title: Bupropion in the Treatment of Methamphetamine Dependence
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: University of Nebraska (Other)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Treatment
Other Study IDs: 0260-07-FB
Record Dates: First submitted 2007-12-11; First posted 2007-12-12 (Estimated); Results first posted 2019-07-26 (Actual); Last update posted 2023-10-10 (Actual); Status verified 2023-09

CONDITIONS: Methamphetamine Use Disorder
Keywords: Methamphetamine; Bupropion SR (Sustained Release)

STUDY DESIGN:
Oversight: Data Monitoring Committee: Yes

ARMS (2):
- Receiving Bupropion SR (Experimental): receiving bupropion SR 12 week course of bupropion SR 150 mg, BID (twice a day)
  Interventions: Drug: bupropion SR
- Treatment as Usual (No Intervention): Not receiving bupropion

INTERVENTIONS:
Drug: bupropion SR — 12 week course of bupropion SR 150 mg, BID
  Arms: Receiving Bupropion SR

SUMMARY:
Methamphetamine dependence is a significant drug use disorder in the Midwest. While a number of psychosocial and pharmacological treatments have been studied, no specific treatments for methamphetamine have been identified. This study is a collaborative pre-clinical and clinical partnership examining bupropion in the treatment of methamphetamine dependence.

DETAILED DESCRIPTION:
Nearly 40% of adults seeking substance use disorders (SUD) treatment in Nebraska report methamphetamine is their drug of choice. In preliminary studies examining bupropion in methamphetamine use, it was well tolerated, reduced craving for methamphetamine and reduced methamphetamine related euphoria. Investigators at the University of Nebraska Medical Center and the University of Nebraska-Lincoln have initiated studies examining bupropion in animals and humans as a potential intervention in addictive disorders. Pre-clinical studies in the Co-Investigator's laboratory were the first to demonstrate the potential utility of bupropion as a pharmacotherapy for methamphetamine use disorders (MUD) while the Principal Investigator studied bupropion as a smoking cessation aid in alcoholics.

The primary goal of this study is to establish an interdisciplinary and translational collaboration to test bupropion in persons in treatment for methamphetamine dependence and to inform pre-clinical studies so as to enhance their practical applicability to clinical settings. The pilot clinical study will examine the treatment effect and safety of a 12 week course of bupropion in persons with methamphetamine use disorder. Concurrently, we will examine the efficacy of bupropion on methamphetamine self-administration in animal models which better simulates clinical approaches.

ELIGIBILITY:
Inclusion Criteria:

* patient in the substance use disorder program at either the Omaha VA Medical Center or at Catholic Charities Campus for Hope
* diagnosis of methamphetamine dependence as well as presence or history of psychosis based on the Diagnostic and Statistical Manual of Mental Disorders Fourth Edition (DSM-IV) criteria (not to include patients in full sustained remission)
* provide names, addresses, and phone numbers of at least two collateral informants who can provide information on their methamphetamine and other drug use during follow-up
* must sign an informed consent as approved by the UNMC Internal Review Board (IRB) and Catholic Charities Research Committee.

Exclusion Criteria:

* a history of severe injury to their brain
* advanced cardiac, pulmonary, renal or liver disease
* predisposition to seizures
* history of bulimia or anorexia nervosa
* current diagnosis of major depressive disorder
* diagnosis or past history of panic disorders, schizophrenia, or bipolar affective disorder
* family history or childhood history of epilepsy or seizures
* history of strokes, brain tumors, or bleeding in the brain.
* used any psychoactive drug within one week of study entry (two weeks for MAO (monoamine oxidase) inhibitors or protriptyline, four weeks for fluoxetine)
* currently using any theophylline product (e.g. Theodur)
* used an investigational drug in any study within the past four weeks
* used a therapeutic course of bupropion SR for > 1 week at any time in the past 12 months or have been evaluated in previous studies examining bupropion SR at anytime
* If female, the participant must not be pregnant or breast feeding

Min Age: 19 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 40 (Actual)
Dates: Start 2007-08-31 (Actual); Primary Completion 2010-04-06 (Actual); Study Completion 2011-05-20 (Actual)

CONTACTS AND LOCATIONS:
Overall Officials: Kathleen M Grant, MD, Principal Investigator — Veterans Affairs Medical Center, Omaha
Locations (2):
- United States (2):
  - Catholic Charities Campus for Hope, Omaha, Nebraska
  - Veterans Affairs Medical Center, Omaha, Omaha, Nebraska

RESULTS

PARTICIPANT FLOW:
Recruitment Details: Dates of recruitment: August 31, 2007 - April 6, 2010 Recruitment from residential substance use disorder treatment programs in Omaha and Lincoln, Nebraska.
Pre-assignment Details: Initially participants were assigned to one of two randomization pools: one group with and one group without psychoses. However as of January 30, 2009 no participants met criteria for randomization to the psychosis arm of the study and the protocol was changed to remove the psychosis randomization pool.
Groups:
- Receiving Bupropion (Sustain Release) SR: receiving bupropion SR
  bupropion SR: 12 week course of bupropion SR 150 mg, (twice a day) BID
Period: Overall Study
Arm/Group | Receiving Bupropion (Sustain Release) SR | Treatment as Usual
Started | 19 | 21
Completed | 18 | 16
Not Completed | 1 | 5

BASELINE CHARACTERISTICS:
Groups:
- Receiving Bupropion SR: receiving bupropion SR
  bupropion SR: 12 week course of bupropion SR 150 mg, BID
- Total: Total of all reporting groups
Arm/Group | Receiving Bupropion SR | Treatment as Usual | Total
Number analyzed (Participants) | 19 | 21 | 40
Age, Continuous [Mean (Standard Deviation); unit: years] | 34 (10.9) | 34 (7.7) | 34 (9.3)
Sex: Female, Male [Count of Participants; unit: Participants]
  Female | 11 | 10 | 21
  Male | 8 | 11 | 19

OUTCOME MEASURES:

1. Primary Outcome: Estimate the Treatment Effect of Bupropion for Methamphetamine (Meth) Dependence.
Description: The primary outcome measure was number of days methamphetamine use/week at weeks 12 and week 24.
Time Frame: Assessed Methamphetamine use at weeks 12 and 24, week 24 reported
Population: Analyses were per protocol and based on number of participants enrolled in study who were not withdrawn from the study.
Measure: Mean (Standard Deviation); unit: days
Groups:
- Receiving Bupropion SR: receiving bupropion SR 12 week course of bupropion SR 150 mg, BID
  bupropion SR: 12 week course of bupropion SR 150 mg, BID
Arm/Group | Receiving Bupropion SR | Treatment as Usual
Number analyzed (Participants) | 19 | 21
days | 5.6 (1.9) | 6.0 (1.3)

ADVERSE EVENTS:
Arm/Group | Receiving Bupropion SR | Treatment as Usual
All-Cause Mortality (participants affected / at risk) | 0/18 | 0/16
Serious Adverse Events (participants affected / at risk) | 0/18 | 0/16
Other Adverse Events (participants affected / at risk) | 0/18 | 0/16

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: No; Agreement restricts PI disclosure of results: No